CLINICAL TRIAL: NCT05637372
Title: Complicated Relationships Between Anterior and Condylar Guidance and Their Clinical Implications- Comparison by Cone Beam Computed Tomography and Electronic Axiography - an Observational Cohort Cross-sectional Study.
Brief Title: Relationships Between Anterior and Condylar Guidance - Comparison by CBCT and Electronic Axiography
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Agata Żółtowska, Doctor, Medical University of Gdansk
Other Study IDs: NKBBN/1043/2021-2022-SCGA
Record Dates: First submitted 2022-11-15; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Temporomandibular Joint Disorders; Occlusion
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients without any disorders and diseases in age range ensuring full temporomandibular joint development.
  Interventions: Radiation: CBCT

INTERVENTIONS:
Radiation: CBCT — CBCT scan

SUMMARY:
The aim of the following study was to investigate the existence of a statistically significant correlation between the incisal features (incisal guidance angle, interincisal angle, overbite, overjet), temporomandibular joint (TMJ) morphology and its function. The hypothesis was:

I. The protrusive movement of the mandible does correlate with the TMJ anatomy. II. The protrusive movement of the mandible does not correlate with the incisal features.

III. The position and relationship of upper and lower permanent incisors do not have a direct and significant effect on the TMJ morphology in young adults.

DETAILED DESCRIPTION:
The study was based on anatomical and functional measurements of the parameters within the masticatory system. The study group was composed in a way that all the participants (age 20-24) had the temporomandibular joints fully developed and at the same time not yet modified by adaptive processes.

ELIGIBILITY:
Inclusion Criteria:

* 20-24 years old

Exclusion Criteria:

* history of trauma, orthodontic treatment or temporomandibular disorders

Ages: 20 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Sagittal condylar guidance angle during protrusion | evaluated within 24h from baseline visit
  recorded with axiograph
Vertical height of the temporomandibular joint fossa | evaluated within 24h from baseline visit
  measured on Cone Beam Computed Tomography
Sagittal condylar guidance angle on Cone Beam Computed Tomography | evaluated within 24h from baseline visit
  conducted in 4 variants of measurements
Features of the incisors | evaluated within 24h from baseline visit
  incisal guidance angle, interincisal angle, overjet, overbite measured on Cone Beam Computed Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Lassmann, DDS, Study Director — Dental Sense Medicover, 80-283 Gdańsk, Poland
Locations (1):
- Dental Sense Medicover, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad KD, Shah N, Hegde C. A clinico-radiographic analysis of sagittal condylar guidance determined by protrusive interocclusal registration and panoramic radiographic images in humans. Contemp Clin Dent. 2012 Oct;3(4):383-7. doi: 10.4103/0976-237X.107419. PMID 23633793
- [Background] Shreshta P, Jain V, Bhalla A, Pruthi G. A comparative study to measure the condylar guidance by the radiographic and clinical methods. J Adv Prosthodont. 2012 Aug;4(3):153-7. doi: 10.4047/jap.2012.4.3.153. Epub 2012 Aug 28. PMID 22977723
- [Background] Dawson PE. Determining the determinants of occlusion. Int J Periodontics Restorative Dent. 1983;3(6):8-21. No abstract available. PMID 6584415
- [Background] Han S, Shin SM, Choi YS, Kim SY, Ko CC, Kim YI. Morphometric analysis for evaluating the relation between incisal guidance angle, occlusal plane angle, and functional temporomandibular joint shape variation. Acta Odontol Scand. 2018 May;76(4):287-293. doi: 10.1080/00016357.2017.1420227. Epub 2018 Jan 11. PMID 29322857
- [Background] Luca, L.; Manfredini, D.; Arveda, N.; Rossi, L.; Siciliani, G. A Cone-Beam Computerized Tomography Assessment of the Relationship between Upper Incisors Inclination and Articular Eminence Features in Orthodontically Untreated Patients with Different Facial Type. J World Fed Orthod 2016, 5 (2), 56-63. https://doi.org/10.1016/j.ejwf.2016.05.001
- [Background] Manfredini D, Lombardo L, Siciliani G. Temporomandibular disorders and dental occlusion. A systematic review of association studies: end of an era? J Oral Rehabil. 2017 Nov;44(11):908-923. doi: 10.1111/joor.12531. Epub 2017 Jul 2. PMID 28600812